CLINICAL TRIAL: NCT01384617
Title: Roux-en-Y Anastomosis of the Pancreatic Stump Following Distal Pancreatectomy
Brief Title: Trial Assessing Roux-en-Y Anastomosis of the Pancreatic Stump to Prevent Pancreatic Fistula Following Distal Pancreatectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wakayama Medical University (Other)
Collaborators: Osaka University (Other); Nara Medical University (Other); Kyoto Prefectural University of Medicine (Other); Kansai Rosai Hospital (Other); Hyogo Medical University (Other)
Responsible Party: Principal Investigator, Hiroki Yamaue, Second Department of Surgery, Wakayama Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KNOW study-1101
Record Dates: First submitted 2011-06-22; First posted 2011-06-29 (Estimated); Last update posted 2016-07-21 (Estimated); Status verified 2016-07

CONDITIONS: Pancreatic Cancer; Pancreatic Cystic Lesions; Chronic Pancreatitis; Pancreatic Neuroendocrine Tumors; Pancreatic Pseudocysts
Keywords: distal pancreatectomy; pancreatic fistula; pancreaticojejunostomy; Roux-en-Y anastomosis; stapling closure
MeSH Terms: conditions — Pancreatic Neoplasms; Pancreatitis, Chronic; Pancreatic Pseudocyst; Pancreatic Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Roux-en-Y anastomosis of the pancreatic stump (Experimental): end-to-side pancreaticojejunostomy into a retrocolic Roux-en-Y reconstruction. The pancreaticojejunostomy anastomosis is performed in duct-to-mucosa.
  Interventions: Procedure: Roux-en-Y anastomosis of the pancreatic stump
- Stapling closure of the pancreatic stump (Active Comparator): Echelon 60 with a gold cartridge provide provides precise and uniform wide compression throughout the entire 60mm length with compressible thickness to 1.8mm, which can attach two triple-staggered rows of titanium staples.
  Interventions: Procedure: Stapling closure of the pancreatic stump

INTERVENTIONS:
Procedure: Stapling closure of the pancreatic stump — Echelon 60 with a gold cartridge provide provides precise and uniform wide compression throughout the entire 60mm length with compressible thickness to 1.8mm, which can attach two triple-staggered rows of titanium staples.
  Arms: Stapling closure of the pancreatic stump
Procedure: Roux-en-Y anastomosis of the pancreatic stump — end-to-side pancreaticojejunostomy into a retrocolic Roux-en-Y reconstruction. The pancreaticojejunostomy anastomosis is performed in duct-to-mucosa.
  Arms: Roux-en-Y anastomosis of the pancreatic stump

SUMMARY:
The objective is to clarify Roux-en-Y anastomosis of the pancreatic stump decreases pancreatic fistula following distal pancreatectomy, compared with stapling closure of the pancreatic stump.

DETAILED DESCRIPTION:
The objective of this study was to clarify Roux-en-Y anastomosis of the pancreatic stump prevents pancreatic fistula after distal pancreatectomy (DP) compared to stapling closure of the pancreatic stump in a prospective randomized controlled trail.

Various methods and technique for treating surgical stump of the remnant pancreas have been reported to reduce pancreatic fistula after DP. However, appropriate surgical stump closure after DP is still controversial.

The primary endpoint in this trial was defined as the incidence of pancreatic fistula .

ELIGIBILITY:
Inclusion Criteria:

1. disease of pancreatic body and tail
2. PS (ECOG Performance Status Scale):0-1
3. Age: 20 years or older
4. distant metastases are not diagnosed preoperatively. Eligible for this clinical study when only distal pancreatectomy contributes to the favorable prognosis even if patients with pancreatic neuroendocrine cancer have the liver metastasis.
5. Adequate organ functions filled the following criteria within two weeks from enrollment:

1.White blood cell： >3,500/mm3 or <12,000/mm3 2.Neutrophilic leukocyte >2,000/mm3 3.Platelet>100,000/mm3 4.Hemoglobin > 9.0g/dL 5.Total bilirubin <2.0mg/dL 6.AST and ALT<150IU/L 7.Creatinine <1.5mg/dL 6)Patients who can provide written informed consent

Exclusion Criteria:

1. Patients with severe liver cirrhosis or active hepatitis
2. Patients with respiratory illness that requires oxygen administration
3. .Patients with chronic renal failure requiring dialysis
4. Patients with active duplicative malignant disease affecting adverse event
5. Others, patients who are unfit for the study as determined by the attending physician

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2011-06; Primary Completion 2014-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Incidence of pancreatic fistula defined by ISGPF classification | 3 month after operation

SECONDARY OUTCOMES:
morbidity | 3 months after opeartion
postoperative hospital stay | 3 month after operation
quality of life | 2 years after operation
new onset or worsening diabetes | 2 years after opeartion
nutritional status | 2 years after opeartion
mortality | 3 months after operation
Incidence of pancreatic fistula gradeB/C defined by ISGPF classification | 3 months after oepration
Incidence of pancreatic fistula grade B/C stratified based on thickness of pancreas parenchyma | 3 months after oepration
Incidence of pancreatic fistula stratified based on thickness of pancreas parenchyma | 3 months after operation

CONTACTS AND LOCATIONS:
Overall Officials: Manabu Kawai, MD, Principal Investigator — Wakayama Medical University, School of Medicine
Locations (1):
- Second Department of Surgery, Wakayama Medical University, School of Medicine, Wakayama, Japan

REFERENCES:
- [Background] Olah A, Issekutz A, Belagyi T, Hajdu N, Romics L Jr. Randomized clinical trial of techniques for closure of the pancreatic remnant following distal pancreatectomy. Br J Surg. 2009 Jun;96(6):602-7. doi: 10.1002/bjs.6620. PMID 19434697
- [Background] Kleeff J, Diener MK, Z'graggen K, Hinz U, Wagner M, Bachmann J, Zehetner J, Muller MW, Friess H, Buchler MW. Distal pancreatectomy: risk factors for surgical failure in 302 consecutive cases. Ann Surg. 2007 Apr;245(4):573-82. doi: 10.1097/01.sla.0000251438.43135.fb. PMID 17414606
- [Background] Wagner M, Gloor B, Ambuhl M, Worni M, Lutz JA, Angst E, Candinas D. Roux-en-Y drainage of the pancreatic stump decreases pancreatic fistula after distal pancreatic resection. J Gastrointest Surg. 2007 Mar;11(3):303-8. doi: 10.1007/s11605-007-0094-2. PMID 17458602
- [Background] Knaebel HP, Diener MK, Wente MN, Buchler MW, Seiler CM. Systematic review and meta-analysis of technique for closure of the pancreatic remnant after distal pancreatectomy. Br J Surg. 2005 May;92(5):539-46. doi: 10.1002/bjs.5000. PMID 15852419
- [Result] Diener MK, Seiler CM, Rossion I, Kleeff J, Glanemann M, Butturini G, Tomazic A, Bruns CJ, Busch OR, Farkas S, Belyaev O, Neoptolemos JP, Halloran C, Keck T, Niedergethmann M, Gellert K, Witzigmann H, Kollmar O, Langer P, Steger U, Neudecker J, Berrevoet F, Ganzera S, Heiss MM, Luntz SP, Bruckner T, Kieser M, Buchler MW. Efficacy of stapler versus hand-sewn closure after distal pancreatectomy (DISPACT): a randomised, controlled multicentre trial. Lancet. 2011 Apr 30;377(9776):1514-22. doi: 10.1016/S0140-6736(11)60237-7. PMID 21529927
- [Result] Zhou W, Lv R, Wang X, Mou Y, Cai X, Herr I. Stapler vs suture closure of pancreatic remnant after distal pancreatectomy: a meta-analysis. Am J Surg. 2010 Oct;200(4):529-36. doi: 10.1016/j.amjsurg.2009.12.022. Epub 2010 Jun 9. PMID 20538249
- [Result] Bassi C, Dervenis C, Butturini G, Fingerhut A, Yeo C, Izbicki J, Neoptolemos J, Sarr M, Traverso W, Buchler M; International Study Group on Pancreatic Fistula Definition. Postoperative pancreatic fistula: an international study group (ISGPF) definition. Surgery. 2005 Jul;138(1):8-13. doi: 10.1016/j.surg.2005.05.001. PMID 16003309
- [Derived] Kawai M, Hirono S, Okada K, Sho M, Nakajima Y, Eguchi H, Nagano H, Ikoma H, Morimura R, Takeda Y, Nakahira S, Suzumura K, Fujimoto J, Yamaue H. Randomized Controlled Trial of Pancreaticojejunostomy versus Stapler Closure of the Pancreatic Stump During Distal Pancreatectomy to Reduce Pancreatic Fistula. Ann Surg. 2016 Jul;264(1):180-7. doi: 10.1097/SLA.0000000000001395. PMID 26473652
- [Derived] Okada K, Kawai M, Tani M, Hirono S, Miyazawa M, Shimizu A, Kitahata Y, Yamaue H. Isolated Roux-en-Y anastomosis of the pancreatic stump in a duct-to-mucosa fashion in patients with distal pancreatectomy with en-bloc celiac axis resection. J Hepatobiliary Pancreat Sci. 2014 Mar;21(3):193-8. doi: 10.1002/jhbp.16. Epub 2013 Jul 22. PMID 23878017